CLINICAL TRIAL: NCT00088218
Title: Randomized Phase II Study of Clofarabine Alone Versus Clofarabine in Combination With Low-Dose Cytarabine in Previously Untreated Patients >= 60 Years With AML and High-Risk MDS
Brief Title: Clofarabine vs Clofarabine in Plus With Low-Dose Ara-C in Previously Untreated Patients With Acute Myeloid Leukemia (AML) and High-Risk Myelodysplastic Syndromes (MDS).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2004-0183
Record Dates: First submitted 2004-07-22; First posted 2004-07-23 (Estimated); Results first posted 2011-05-09 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2011-04

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: Acute Myeloid Leukemia; AML; High-Risk Myelodysplastic Syndrome; MDS; Clofarabine; Cytarabine; ara-C
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Clofarabine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clofarabine (Active Comparator): Clofarabine intravenous (IV) 30 mg/m^2 daily times 5 days
  Interventions: Drug: Clofarabine
- Clofarabine Plus Ara-C (Active Comparator): Clofarabine IV 30 mg/m^2 daily times 5 days + Ara-C 20 mg/m^2 subcutaneously daily times 14 days.
  Interventions: Drug: Clofarabine; Drug: Ara-C

INTERVENTIONS:
Drug: Clofarabine — 1-hour IV infusion 30 mg/m^2 daily times 5 days (Days 1-5)
  Other Names: Clolar; Clofarex
Drug: Ara-C — 20 mg/m^2 subcutaneously daily times 14 days (Days 1-14). On Days 1 to 5 of each course, clofarabine will precede injection of ara-C by approximately 4 hours (+/- 1 hour).
  Other Names: Cytarabine; Cytosar; DepoCyt; Cytosine arabinosine hydrocloride
  Arms: Clofarabine Plus Ara-C

SUMMARY:
The goal of this clinical research study is to study how effective treatments with clofarabine alone and clofarabine given in combination with ara-C are in the treatment of leukemia and high-risk myelodysplastic syndrome (MDS) in patients who are 60 years or older. The safety of these treatments will also be compared.

DETAILED DESCRIPTION:
Clofarabine is a chemotherapy drug that is designed to interfere with the growth and development of cancer cells. Ara-C is a chemotherapy drug which is approved for the treatment of AML and MDS. Although there is experience with the combination of both drugs, there have not been trials that explored the particular doses and schedule of clofarabine plus ara-C that you may receive.

Before you can start treatment on the study, you will have what are called "screening tests". These tests will help the doctor decide if you are eligible to take part in the study. You will have a complete medical history and physical exam. You will also be asked about what medications you are taking currently and about the level of your daily activities. About 2 tablespoons of blood will be collected for routine blood tests and to make sure you are not at increased risk for developing side effects.

Before your first treatment (usually within 14 days), you may have bone marrow samples collected. To collect a bone marrow sample, an area of the hip or chest bone is numbed with anesthetic and a small amount of bone marrow is withdrawn through a large needle. The procedure will be explained to you by your doctor and will require you to sign a separate consent document.

Early study results showed that there is clearly a better response with the combination treatment compared to the clofarabine alone treatment. Because of this, all participants in this study will now be assigned to the clofarabine plus ara-C group. You will receive clofarabine through a vein daily for 5 days in a row. In addition, you will receive injections of ara-C under the skin once a day for 14 days in a row. On those days when both clofarabine and ara-C are taken, the clofarabine will be given approximately 4 hours before the ara-C injections. You can be taught to give the ara-C injections to yourself. Each cycle may be repeated every 3 to 6 weeks. You will be required to record the injections in a medication diary.

Up to 2 of these cycles (for both groups) can be given at this dose schedule. If you show a response to treatment, you can continue with up to 12 cycles of therapy, during which clofarabine will be given for 3 days instead of 5 and ara-C for 7 days instead of 14. Maintenance courses may be given on average every 4 to 7 weeks.

Before every treatment course, you will have a physical exam including measurement of your weight and vital signs. You will also be asked how you are feeling and how you are able to go about your daily routine. At least once a week (more often if your doctor feels it is necessary), you will have blood samples (about 1-2 teaspoons) collected for routine lab tests. Around 3 weeks after your first treatment, you may have samples of bone marrow collected. After that, the bone marrow collections will be performed every 2 weeks (or more often if your doctor feels it is necessary). The bone marrow sample will be tested to evaluate the response of the disease to therapy.

You will need to stay in Houston for the first 4 weeks of treatment. After that, you have to return to Houston to receive the clofarabine treatment, but you can have check-up visits and blood tests with your local doctor. If the disease gets worse or you experience any intolerable side effects, you will be taken off the study and your doctor will discuss other treatment options with you.

After you finished your treatment, and as long you are participating on this study you will be scheduled every 3-6 months to check on the status of the disease and your overall health as long as you stay on the study. Once you are taken off the study, your doctor will decide how often you will have follow-up as part of your standard care.

This is an investigational study. Clofarabine is authorized by the Food and Drug Administration (FDA) for use in research only. Up to 108 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated AML and high-risk MDS ( > 10% blasts, or International Prognostic Scoring System (IPSS) intermediate-2). Prior therapy with hydroxyurea, single agent chemotherapy (e.g. decitabine), hematopoietic growth factors, biological or "targeted" therapies are allowed.
* Age > 60 years.
* Eastern Cooperative Oncology Group (ECOG) performance status </= 2.
* Sign a written informed consent form.
* Adequate liver function (total bilirubin < 2mg/dL,serum glutamic pyruvic transaminase (SGPT) or Serum glutamic oxaloacetic transaminase (SGOT) < x 4 upper limit of normal (ULN)) and renal function (serum creatinine < 2mg/dL).

Exclusion Criteria:

* Patients with >= New York Heart Association (NYHA) grade 3 heart disease as assessed by history and/or physical examination.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2004-07; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Faderl, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Faderl S, Ravandi F, Huang X, Garcia-Manero G, Ferrajoli A, Estrov Z, Borthakur G, Verstovsek S, Thomas DA, Kwari M, Kantarjian HM. A randomized study of clofarabine versus clofarabine plus low-dose cytarabine as front-line therapy for patients aged 60 years and older with acute myeloid leukemia and high-risk myelodysplastic syndrome. Blood. 2008 Sep 1;112(5):1638-45. doi: 10.1182/blood-2007-11-124602. Epub 2008 Jun 18. PMID 18565853
- See also: M.D. Anderson Cancer Center's website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period 7/21/04 - 2/15/08; all patients were registered at The University of Texas M.D. Anderson Cancer Center.
Period: Overall Study
Arm/Group | Clofarabine | Clofarabine Plus Ara-C
Started | 16 | 79
Completed | 16 | 79
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clofarabine | Clofarabine Plus Ara-C | Total
Number analyzed (Participants) | 16 | 79 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 12 | 13
  >=65 years | 15 | 67 | 82
Age Continuous [Median (Full Range); unit: years] | 72 [60 to 83] | 70 [60 to 82] | 70 [60 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 34 | 38
  Male | 12 | 45 | 57
Region of Enrollment [Number; unit: participants]
  United States | 16 | 79 | 95

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response
Description: Participant responses are categorized as 'Complete Remission,' Complete Remission, No Platelet Recovery,' 'No Response.'
  Complete Remission: Disappearance of all clinical and/or radiologic evidence of disease. Neutrophil count > 1.0 x 109/L and platelet count > 100 x 109/L, and normal bone marrow differential (< 5% blasts); Complete Remission, No Platelet Recovery: Peripheral blood and bone marrow results as for CR, but with platelet counts of < 100 x 109/L.
  Blood draws once a week until remission then every 2 to 8 weeks during therapy.
Time Frame: Every 2 to 8 weeks
Population: All treated subjects.
Measure: Number; unit: Participants
Arm/Group | Clofarabine | Clofarabine Plus Ara-C
Number analyzed (Participants) | 16 | 79
Participants
  Complete Remission | 5 | 49
  Complete Remission, No Platelet Recovery | 0 | 4
  No Response | 11 | 26

ADVERSE EVENTS:
Time Frame: 3 years 7 months
Arm/Group | Clofarabine | Clofarabine Plus Ara-C
Serious Adverse Events (participants affected / at risk) | 12/16 | 39/79
Other Adverse Events (participants affected / at risk) | 16/16 | 54/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine (N=16) | Clofarabine Plus Ara-C (N=79)
GI Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 5 (5)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 8 (8)
Adult Respiratiory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 6 (6)
Pneumonia (Infections and infestations) | 2 (2) | 8 (8)
Prolonged Myelosuppression (Blood and lymphatic system disorders) | 1 (1) | 6 (8)
Febrile Neutropenia (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcus Infection (Infections and infestations) | 0 (0) | 2 (2)
Sepsis Infection (Infections and infestations) | 1 (1) | 0 (0)
Sinus Infection (Infections and infestations) | 0 (0) | 1 (1)
Elevated Triponin (Cardiac disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Syncope (General disorders) | 0 (0) | 2 (2)
Infection (Infections and infestations) | 1 (1) | 3 (4)
Fungal Infection (Infections and infestations) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Secondary Malignancy Colon Cancer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bactremia Infection (Infections and infestations) | 0 (0) | 1 (1)
Secondary Malignancy Squamous Cell Carcinoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine (N=16) | Clofarabine Plus Ara-C (N=79)
Diarrhea (Gastrointestinal disorders) | 12 (12) | 48 (48)
Nausea (Gastrointestinal disorders) | 12 (12) | 39 (39)
Hyperbilirubinemia (Hepatobiliary disorders) | 10 (10) | 49 (49)
Mucositis (Gastrointestinal disorders) | 3 (3) | 24 (24)
Elevated alanine aminotransferase (Hepatobiliary disorders) | 10 (10) | 35 (35)
Skin rash (Skin and subcutaneous tissue disorders) | 9 (9) | 37 (37)
Headache (Nervous system disorders) | 6 (6) | 27 (27)
Emesis (Gastrointestinal disorders) | 9 (9) | 27 (27)
Edema (General disorders) | 6 (6) | 29 (29)
Elevated aspartate transaminase (Hepatobiliary disorders) | 5 (5) | 25 (25)
Anorexia (Gastrointestinal disorders) | 3 (3) | 16 (16)
Elevated alkaline phosphatase (Hepatobiliary disorders) | 3 (3) | 15 (15)
Elevated Creatinine (Blood and lymphatic system disorders) | 5 (5) | 14 (14)
Acute renal failure (Renal and urinary disorders) | 2 (2) | 3 (3)
Fatigue (General disorders) | 3 (3) | 9 (9)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 8 (8)
Hand-Foot syndrome (Nervous system disorders) | 2 (2) | 7 (7)
Facial flushing (General disorders) | 1 (1) | 6 (6)
Puritis (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)
Chest tightness (Cardiac disorders) | 0 (0) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No